CLINICAL TRIAL: NCT03424850
Title: A Phase I/II Dose-escalation Study Evaluating the Safety and Efficacy of 21 Gy, 23 Gy and 25 Gy for High Dose Rate (HDR) Prostate Brachytherapy
Brief Title: Safety and Efficacy of 21 Gy, 23 Gy and 25 Gy for High Dose Rate (HDR) Prostate Brachytherapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201801118
Record Dates: First submitted 2018-01-23; First posted 2018-02-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- HDR brachytherapy - 21 Gy (Experimental): -All patients will be treated with a single implant and single HDR fraction. Treatment will be delivered within a single 24-hour period measured from the beginning of the implant procedure. All patients will receive a dose of 21 Gy.
  Interventions: Radiation: HDR brachytherapy
- HDR brachytherapy - 23 Gy (Experimental): -All patients will be treated with a single implant and single HDR fraction. Treatment will be delivered within a single 24-hour period measured from the beginning of the implant procedure. All patients will receive a dose of 23 Gy.
  Interventions: Radiation: HDR brachytherapy
- HDR brachytherapy - 25 Gy (Experimental): -All patients will be treated with a single implant and single HDR fraction. Treatment will be delivered within a single 24-hour period measured from the beginning of the implant procedure. All patients will receive a dose of 25 Gy.
  Interventions: Radiation: HDR brachytherapy

INTERVENTIONS:
Radiation: HDR brachytherapy — * Dose constraints for 21 Gy:
    * Bladder and rectum: V70 < 1 cc
    * Urethra: V115 < 1 cc
    * V135: 0%
  * Dose constraints for 23 Gy:
    * Bladder and rectum: V65 < 1 cc
    * Urethra: V105 < 1 cc
    * V125: 0%
  * Dose constraints for 25 Gy:
    * Prostate V100 >90% (>95% preferred)
    * Bladder and rectum: V70 < 1 cc, Dmax <115%
    * Urethra: V110 < 1 cc, Dmax <120%

SUMMARY:
The purpose of this research study is to learn more about the outcomes and early and late side effects of treating early stage prostate cancer with high dose rate brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of early stage prostate cancer.
* Must be considered either low-risk (T1-T2a, Gleason ≤ 6, PSA < 10 ng/mL) or favorable intermediate-risk (Gleason 3 +4 = 7, percentage of positive biopsy cores < 50%, no more than one NCCN intermediate risk factor).
* Prior androgen deprivation therapy is allowed and may have been initiated up to 6 months prior to the date of the HDR implant. The complete duration of androgen deprivation therapy can range from 4 months to 36 months provided it has been initiated no more than 6 months prior to the date of the HDR implant.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior radiation therapy to the prostate or lower pelvis encompassing the prostate.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only.
* Currently receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Unable to undergo general, spinal or local anesthesia.
* Prior TURP with a sufficiently large defect that would compromise the integrity of the implant per clinician's assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-02-27 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Biochemical control experienced by patients with prostate cancer treated with an HDR implant | Through 3 years after implant
  -Response will be determined by PSA. The Phoenix definition will be used for determining biochemical failure: a rise of 2 ng/mL or more above the PSA nadir

SECONDARY OUTCOMES:
Rate of acute toxicity experienced by patients with prostate cancer treated with an HDR implant | From start of treatment through 90 days
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Rate of late toxicity experienced by patients with prostate cancer treated with an HDR implant | From day 91 through 3 years after implant
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.

OTHER OUTCOMES:
Optimal dose of radiation | Through 3 months after completion of implant for all patients enrolled (estimated to be 5 years and 3 months)
  -The optimal dose is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity within the DLT assessment period (3 months after implant) OR the maximally administered dose if fewer than 2 patients in that cohort experience DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Hiram A Gay, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu